CLINICAL TRIAL: NCT01276444
Title: Comparison of Goal-directed Algorithms of Hemodynamic Therapy After Combined Valve Repair: a Randomized Clinical Trial
Brief Title: Comparison of Goal-directed Algorithms of Hemodynamic Therapy After Combined Valve Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Northern State Medical University, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SCVO2-2008
Record Dates: First submitted 2011-01-04; First posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: Valvular Heart Disease
Keywords: valve repair; postoperative period; goal-directed therapy; pulmonary artery catheter; transpulmonary thermodilution; central venous oxygen saturation
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pulmonary artery catheter (PAC) (Active Comparator): PAC was used to guide hemodynamic therapy after combined valve repair
  Interventions: Device: Swan-Ganz catheter
- COMPLEX (Active Comparator): An combination of transpulmonary thermodilution and continuous monitoring of central venous saturation was used to guide hemodynamic therapy after combined valve repair surgery.
  Interventions: Device: transpulmonary thermodilution + central venous saturation

INTERVENTIONS:
Device: Swan-Ganz catheter — the data s=derived from PAC included pulmonary artery occlusion pressure etc
  Other Names: Not actual
  Arms: Pulmonary artery catheter (PAC)
Device: transpulmonary thermodilution + central venous saturation — Described in details above
  Other Names: Non actual
  Arms: COMPLEX

SUMMARY:
Valvular repair and repair surgery is rapidly progressing yet rather challenging aspect of current cardiosurgical practice.

Several approaches were introduced into the clinical practice to alleviate systemic inflammatory response induced by cardiopulmonary bypass and organ-specific injury including meticulous haemodynamic monitoring, pharmacological heart preconditioning, systemic use of anti-inflammatory agents, prevention of coagulopathy, and induced topical and systemic hypothermia. An in-depth monitoring of haemodynamics, oxygen transport, and vascular permeability is of a great clinical value to control the efficacy of these approaches.

Therefore, the aim of this study was to compare two algorithms of goal-directed therapy aimed to achieve a postoperative haemodynamic optimization in combined valve repair surgery.

DETAILED DESCRIPTION:
Forty-three adult patients scheduled for elective two valve replacement/repair were enrolled into randomised single-centre study. All interventions were performed in cardiosurgical department of City hospital #1 (Arkhangelsk, Russian Federation) by the same surgical team. Three patients were excluded from the analysis; two - due to protocol violation and one - due to inadequate surgical correction diagnosed by intraoperative transoesophageal echocardiography.

Day before surgery patients were asked for informed consent and randomized in two groups. In the first group postoperative haemodynamic optimization was targeted on parameters provided by pulmonary artery catheter (the PAC-group, n = 20): pulmonary arterial occlusion pressure, cardiac index (LifeScope monitor, Nihon Kohden, Japan) and hemoglobin blood level. In the second group haemodynamics was managed using parameters given by transpulmonary thermodilution (the COMPLEX-group), that included cardiac index, global end-diastolic volume index, extravascular lung water index, continuous central venous oxygen saturation, and oxygen delivery index as measured with PiCCO2 monitor (Pulsion Medical Systems, Munich, Germany. In addition, mean arterial pressure, heart rate, and hemoglobin concentration were included into both PAC- and PiCCO2-driven protocols.

ELIGIBILITY:
Inclusion Criteria:

* Two valve repair / replacements
* Age above 18
* Informed consent

Exclusion Criteria:

* pulmonary hypertension
* insulin-dependent diabetes mellitus
* severe atherosclerosis of femoral arteries
* severe respiratory failure
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-01; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Mortality | Day 28
  Mortality rate at Day 28

SECONDARY OUTCOMES:
Fit for discharge | non actual
  Formal 'fit for discharge from ICU' criteria
Vasoactive support | 7 days
  Duration of vasopressor and or inotrope support
Duration of respiratory support | Day 7
  The total duration of the respiratory support

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y. Kirov, MD, PhD, Principal Investigator — Northern State Medical University
Locations (1):
- City hospital # 1 / Northern State Medical University,, Arkhangelsk, Russia